CLINICAL TRIAL: NCT06500117
Title: Digital Mindfulness Training Programme for Smoking Cessation and Maintenance a Mixed-method Pilot Study
Brief Title: Digital Mindfulness Training Programme for Smoking Cessation and Maintenance
Acronym: HowToMind
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DEMINA IReSP/INCa 2023
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Smoking-related Disorder
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patient (Experimental)
  Interventions: Other: eMind application; Other: questionnaires; Other: focus groupe

INTERVENTIONS:
Other: eMind application — learning phase accompanied by application for 8 weeks, then independent practical application phases
Other: questionnaires — Visual Analogue Scale VAS ("craving") and Mobile Application Rating Scale MARS-F
Other: focus groupe — Patients who so wish will be able to give us more detailed feedback on the application. The focus groups will be carried out between visit 3 and visit 4.

SUMMARY:
Although there are several effective medicinal approaches for smoking cessation, relapses are frequent and the proportion of people who remain abstinent is low (around 15-25% 6 months after withdrawal). New approaches are therefore needed to make it easier to stop smoking.

Mindfulness-based interventions (MBIs) are effective in depression, stress reduction and chronic pain (Goldberg et al., 2017, Khoury et al., 2015, Hilton et al., 2017). There is also evidence of efficacy in smoking cessation with a relative risk of 1.88 95% CI [1.04; 3.40] of abstinence at 17 to 24 weeks after MBI (Oikonomou, 2016).

Typically, MBIs take the form of 8-week programmes with weekly group sessions. However, many patients are not able to attend a full 8-week programme. In addition, these programmes are only accessible to a small number of patients due to the lack of trained professionals and the out-of-pocket costs.

In response to these limitations, smartphone applications have been developed and evaluated, but none has been shown to be effective in smoking cessation. What's more, none of the evaluated applications offered the equivalent of a conventional 8-week MBI.

Furthermore, it has now been demonstrated in the international literature that involving patients, service users and relatives in the development and conduct of health research projects has become a means of achieving effective, high-quality integration of healthcare (Fusco, 2020) as well as improving the overall quality of health research (Shen, 2017). When PUPs are involved not as research subjects but as research partners in the health research process, this can lead to "significant changes in outcomes for patients and health systems, and the realignment of research processes and outcomes to be patient-centred" (Bird, 2020).

The involvement of PUPs has become a requirement of many funding programmes and journals, as well as an international health policy priority.

We are therefore developing an eMind application - the first electronic MBI for smoking cessation that allows patients to follow a complete 8-week programme and that recreates the conditions of a classic MBI as closely as possible. The application will be available on the EXOLIS platform. This platform is offered by the Agence Régionale de Santé Bourgogne - Franche Comté in partnership with GRADeS (Groupement Régional d'Appui au Développement de la eSanté).

The eMind application will be co-constructed: it will be based on a research partnership involving patients. An initial version of the content has been created in the university hospital addictionology department by healthcare professionals trained in mindfulness. This first version of the application - a beta version - will be modified according to the feedback received from patients. To reward their contribution to the final version of the application, patients will be compensated in the form of a gift card. Once the changes have been taken into account, a feedback session will be organised to present the results of the study and the new version of eMind.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent
* Adult aged 18 and over
* Smoker with a smoking-related disorder according to DSM-5 criteria
* Motivated to stop smoking
* With daily access to a smartphone
* Able to understand spoken and written French

Exclusion Criteria:

* Person subject to a legal protection measure (curatorship, guardianship)
* Persons under court order
* People with cognitive problems that prevent mindfulness training
* Currently using other smoking cessation treatments (burpropion, varenicline) except NRT
* suffering from an acute psychiatric or somatic disorder requiring hospitalisation / not stabilised
* With a contraindication to nicotine replacement therapy
* With an alcohol use disorder or using illicit substances
* Anyone who is pregnant, breastfeeding or planning to become pregnant in the next 6 months
* Not affiliated to national health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The acceptability of the beta version of eMind will be assessed by how regularly it is used. | Usability will be assessed after 8 weeks' use of the application.
  Based on the rhythm of the videos and audio provided by the application, we will define people who use eMind at least 4 times a week for 8 weeks as active users, those who use the application 1 to 3 times a week as occasional users, and those who no longer use the application after 8 weeks as users who have given up using the application.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demina A, Soudry-Faure A, Petit B, Meunier-Beillard N, Trojak B. Usability of a digital mindfulness training program for smoking cessation: A mixed-method single-center pilot study protocol (HowToMind). PLoS One. 2025 Feb 20;20(2):e0318686. doi: 10.1371/journal.pone.0318686. eCollection 2025. PMID 39977412